CLINICAL TRIAL: NCT06671951
Title: Effectiveness of Focal Vibration in Enhancing Lower Extremity Speed and Power in Athletes
Brief Title: Focal Vibration for Enhancing Athletic Speed and Ppower
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Maxim Canet Vintró, Msc, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CBAS-2023-05
Record Dates: First submitted 2024-07-25; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: To Assess the Effectiveness of a Focal Vibration Treatment on Squat Power and Speed in Athletes Who Perform Squats

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibration group (Experimental): The vibration group receives an intervention with focal vibration heads from Wintecare on the rectus femoris, vastus lateralis and vastus medialis , at the same time that the athelte is doing active muscle contractions.
  Interventions: Other: Focal Vibration
- Sham group (Sham Comparator): The placebo group receives the same protocol but the head of the focal vibration machine is not in contact with the patient's skin.
  Interventions: Other: Sham focal vibration

INTERVENTIONS:
Other: Focal Vibration — Focal vibration is a 3x3 electrode placed on the athlete's muscle belly, and emits a high frequency vibration (150Hz) to stimulate the muscle spindle and generate greater muscle activation.
  Other Names: Local Vibration
  Arms: Vibration group
Other: Sham focal vibration — Is a focal vibration intervention but without conctact in the athelte's skin. Doing this we got a sham therapy
  Arms: Sham group

SUMMARY:
A focal vibration device will be used to perform an activation and warm-up protocol before performing a set of 7 repetitions of squat with 60% of your 1RM.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must have signed the informed consent form to assess their inclusion in the study.
* Familiarity with the technique and practice of the weighted free squat.
* Training at least 3 times per week.

Exclusion Criteria:

* Volunteers who have suffered a sports injury during the last two months or are unable to perform physical activity.
* Have previously received an intervention with focal vibration.
* Not understanding the information provided by the therapist.
* Participate in other research studies.
* Be undergoing pharmacological medical treatment that may interfere with the measurements, such as treatment with anticonvulsants, antidepressants, etc.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-06 (Estimated)

PRIMARY OUTCOMES:
Mean Speed during squat | 1 minute
  A linear transducer (Vitruve VBT) was used to measure the mean speed during the squat. The tether device was attached to the right side of the barbell around the widest part of the collar on the inside and this converts the subject's movement with the barbell into an electrical signal that will record the mean speed and of the exercise. Subjects will per-form 7 repetitions at 0,85 m/s at the maximum possible speed with the optimal load to generate the maximum power.
  Linear transducers which have greater accuracy (5%) and reliability (ICC: 0.752; 95% CI: 0.548 - 0.855) compared to other devices in terms of velocity-based training (VBT) meas-urement.
Mean Power during squat | 1 minute
  A linear transducer (Vitruve VBT) was used to measure the mean power during the squat. The tether device was attached to the right side of the barbell around the widest part of the collar on the inside and this converts the subject's movement with the barbell into an electrical signal that will record the mean power of the exercise. Subjects will per-form 7 repetitions at 0,85 m/s at the maximum possible speed with the optimal load to generate the maximum power.
  Linear transducers which have greater accuracy (5%) and reliability (ICC: 0.752; 95% CI: 0.548 - 0.855) compared to other devices in terms of velocity-based training (VBT) meas-urement.

SECONDARY OUTCOMES:
Scale of perceived effort during squat | 1 minute
  Just after the end of the series of 7 repetitions the sensation of effort perceived by the athlete was measured with the modified BORG scale (0-10), being 0 the lowest perceived effort and 10 being the highest effort.
Participant's rating of clinical change. Global Rating of Change Scale (GROC scale). | 1 minute
  At the end of the free bar squat after the warm-up and the intervention, the subject will be asked if he/she has felt improvement or worsening between the first time and the last time he/she performed the test. The participant's rating of clinical change will be evaluated with a Global Rating of Change Scale (GROC scale). This is a scale of 15 items, of which +7 are improvement and -7 are deterioration, and with 1 central item with no clinical change. Values from the fourth item of improvement or deterioration will be considered clinically significant, values between the three item of improvement and the three item of deterioration will be considered as no clinically significant changes. The test-retest reliability has proven to be good (ICC 0.90).
Muscle Activity | 1 minute
  Surface electromyography was used to evaluate the muscle activity of back and lower limb the during squatting task. The muscles assessed were vastus medialis, vastus lateralis, rectus femoris, biceps femoris, gluteus maximus and erector spinae longissimus. Data were obtained for the dominant limb defined as the one preferred to kick a ball.
  the tool to be used is The mDurance® system (mDurance Solutions SL, Granada, Spain). The RMS was the principal variable recorded for muscle activity, expressed as % of MVIC (%MVIC).

IPD SHARING:
Plan to Share IPD: Undecided